CLINICAL TRIAL: NCT05271526
Title: A Multicenter, Single Arm, Non-interventional, Observational, Prospective Study to Assess Demographic Characteristics, Burden of Disease and Short-term Patient Reported Outcomes on Symptom Relief in Severe Eosinophilic Asthma Patients Aged Older Than 18 Qualifying for Treatment With Benralizumab in Russia
Brief Title: Real World Evidence of Benralizumab in Eosinophilic Severe AsThma in Russia (BEST)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00101
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Benralizumab is a humanised, afucosylated, monoclonal antibody against the interleukin (IL)-5 receptor (IL-5R) α subunit that induces direct, rapid, and near-complete depletion of eosinophils in blood, airway tissue, and bone marrow through enhanced antibody-dependent cell-mediated cytotoxicity (ADCC). This apoptotic process involves natural killer cells responsible for the controlled eosinophilic elimination. In the two pivotal phase III trials SIROCCO and CALIMA, benralizumab was well tolerated, significantly reduced asthma exacerbations by up to 51%, and improved lung function as well as disease control in patients with severe, uncontrolled asthma and blood eosinophil count of ≥ 300 cells/μL blood, receiving both ICS and LABA.

According to the summary of product's characteristics (SmPC) of benralizumab in Russia, it can be used for an add-on maintenance treatment for adult patients with severe eosinophilic asthma. All patients enrolled in the BEST study will comply with the SmPC approved by the Russian Ministry of Health.

DETAILED DESCRIPTION:
This is a multicentre, single arm, non-interventional observational, prospective study that will include patients older than 18 years, who qualify for the treatment with benralizumab according to the SmPC in participating research centres (study cites) focusing on severe eosinophilic asthma in Russia. The decision by the physician to start benralizumab is made independently from study inclusion and patient informed consent. Patients who meet the study criteria will be enrolled and, as outlined in the current label of benralizumab approved by Russian Ministry of Health, are planned to receive 3 subcutaneously (s.c.) applied doses of 30 mg benralizumab, from weeks 0 (baseline) every 4 weeks and then every 8 week. A follow-up visit to assess the sustainability of achieved changes will be done after 56 weeks. No study drug will be provided, all patients will be on commercially available drug. Additional two study visits at week 1 and 2 can also be done remotely via phone calls to obtain the paper-based SGRQ, ACQ-5, PGI-C and PGI-S questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Subject eligible for enrolment in the study and treatment for benralizumab according to the specific Russian label and in line with reimbursement condition must meet all the following criteria:

* Male or female patients older than 18 years with physician's confirmed diagnosis of severe, uncontrolled asthma.
* Asthma requiring high-dose ICS plus LABA as maintenance treatment.
* Minimum of 2 exacerbations in the last 12 months. Or 1 exacerbation in case that patient had been receiving oral glucocorticoid therapy for at least 6 continuous months directly before enrollment (equivalent to a prednisolone or prednisone dose of 7.5 to 40.0 mg per day)
* Documented peripheral blood eosinophil count ≥ 300 cells/μL or ≥150 cells/μL blood in case that patient had been receiving oral glucocorticoid therapy for at least 6 continuous months directly before enrollment (equivalent to a prednisolone or prednisone dose of 7.5 to 40.0 mg per day).
* Provision of signed written ICF indicating that they understand the purpose of the study and procedures required for participation in the study.
* Patients must be able and willing to read and comprehend written instructions and comprehend and complete the questionnaires required by the protocol (SGRQ, ACQ-5, PGIC and PGIS).

Exclusion Criteria:

Patients who have previously received benralizumab prior to the start of the study.

* Documented lung diseases other than asthma, e.g. COPD, and not within reimbursed label, e.g pregnancy or lactation.
* Concomitant treatment with any other biologic for any indication or previous treatment with biology. Acceptable wash-out periods for other asthma biologics: ≥4 month or duration of 5 half-lives from last dose of previous biologic. We choose what is longer the 5 half-life or 4 months.
* Currently enrolled in an interventional clinical study in parallel, except:

  * Patients being in parallel documented in a national asthma registry.
  * Patients having completed any other clinical trial including those with biologic treatment ≥4 month or duration of 5 half-lives from last dose of previous biologic. We choose what is longer the 5 half-life or 4 months.
* An acute or chronic condition that, in the investigator's opinion, would limit the patients' ability to complete questionnaires or participate in this study or impact the interpretations of results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit 59 male and female patients aged ≥ 18 years with severe, eosinophilic asthma who meet all inclusion criteria and none of the exclusion criteria (15% drop out). Approximately 10 centers across Russia will participate in the study. Only those centres that have experience with biologic treatment, can initiate treatment with benralizumab and have a good oversight on the severe asthma population (as in some settings the patients are referred for longer term stationary care to achieve asthma control) will be able to participate.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in patient asthma control after initiation of benralizumab in a real-world Russian setting | Up to 6 month
  Mean scores change from baseline in Asthma Control Questionnaire-5 (ACQ-5) after 8 weeks of treatment with benralizumab.
To evaluate the change in respiratory health-related quality of life in a real-world Russian setting | Up to 6 month
  Total scores change from baseline in St. George's Respiratory Questionnaire (SGRQ) after 8 weeks of treatment with benralizumab

CONTACTS AND LOCATIONS:
Locations (1):
- City clinical hospital No57, Moscow, Russia

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00101&attachmentIdentifier=b341e4ce-115f-458d-8739-d53787cb8140&fileName=Study_report_XALOC_synopsis_redacted.pdf&versionIdentifier=